CLINICAL TRIAL: NCT06325293
Title: A Randomized Controlled Non-inferiority Trial of Placebo Versus Macrolide Antibiotics for Mycoplasma Pneumoniae Infection in Children With Community-acquired Pneumonia - the MYTHIC Study
Brief Title: A Trial of Placebo Versus Macrolide for Mycoplasma Pneumoniae Childhood Pneumonia: MYTHIC Study
Acronym: MYTHIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Berger (Other)
Collaborators: SNF Swiss National Foundation (Unknown); Swiss Clinical Trial Organisation (Unknown); SwissPedNet (Unknown)
Responsible Party: Sponsor-Investigator, Christoph Berger, Prof. Dr. med., University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-01295; 207286 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2024-02-26; First posted 2024-03-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-08

CONDITIONS: Community Acquired Pneumonia in Children; Mycoplasma Pneumoniae; Mycoplasma Pneumoniae Pneumonia
Keywords: Mycoplasma pneumoniae; community-acquired pneumonia; randomized controlled trial; Investigator Initiated Clinical Trial (IICT); Paediatric pneumonia; children; placebo; macrolides
MeSH Terms: conditions — Pneumonia, Mycoplasma; Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, multicenter, non-inferiority trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMP arm (Active Comparator): Azithromycin Pfizer® powder for oral suspension:
  1 daily dose for 5 days, 10mg/kg/day on day 1 and 5mg/kg/day on days 2-5
  Interventions: Drug: Azithromycin Pfizer®
- Placebo arm (Placebo Comparator): 5 days of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin Pfizer® — Azithromycin Pfizer® powder for oral suspension will be used in the active comparator arm: 1 daily dose for 5 days, 10mg/kg/day on day 1 and 5mg/kg/day on days 2-5
  Arms: IMP arm
Drug: Placebo — Control comparator arm: 5 days of placebo
  Arms: Placebo arm

SUMMARY:
The goal of this clinical trial is to compare a placebo (a look-alike substance that contains no active drug) with a commonly used antibiotic in children with Mycoplasma pneumoniae (a specific bacterium) induced community-acquired pneumonia. The main question it aims to answer is:

Is antibiotic treatment needed in Mycoplasma pneumoniae (a specific bacterium) induced pneumonia?

Participants will receive either a placebo or a antibiotic treatment and track their symptoms and vital signs until they are healthy.

Researchers will then compare the length of symptoms between the placebo and the antibiotic group.

DETAILED DESCRIPTION:
Mycoplasma pneumoniae (M. pneumoniae) is the most frequently detected bacterial pathogen in community-acquired pneumonia (CAP) in hospitalized U.S. children. Prior to the COVID-19 pandemic, M. pneumoniae was responsible for 8-28% of childhood CAP and thus was substantially contributes to CAP being a leading cause of hospitalization in high-income settings and worldwide morbidity and mortality. After the corona virus disease (COVID)-19 pandemic, M. pneumoniae and its delayed re-emergence remains a thread to children's health. CAP accounts for more treatment days with antibiotics in children's hospitals in the U.S. than any other condition. Macrolides are the first-line treatment for M. pneumoniae infection. Still, there is a lack of evidence for macrolides' the effectiveness in the treatment of M. pneumoniae induced CAP; simultaneously there is an alarmingly increasing antimicrobial resistance among M. pneumoniae. Therefore, childhood CAP, and especially M. pneumoniae, is an important target for antimicrobial stewardship efforts and cost-effectiveness considerations.

The MYTHIC Study is a randomized, double-blind, placebo-controlled, multicenter, non-inferiority trial in 13 Swiss pediatric centers. Previously healthy ambulatory and hospitalized children aged 3-17 years with clinically diagnosed CAP will be screened for a M. pneumoniae infection with Immunoglobulin M (IgM) lateral flow assay. Patients will be randomized 1:1 to receive a 5-day-treatment of macrolides (azithromycin) or placebo.

ELIGIBILITY:
Inclusion criteria for screening phase:

* Children aged 3-17 years (from 3rd up to 18th birthday) presenting to the emergency department (ED) who will be managed ambulatory or will be admitted to general ward.
* Clinical diagnosis of CAP:

  1. Diagnosis defined as the treating physician's documented diagnosis of CAP; AND
  2. Fever ≥38.0°C (measured by any method [i.e., ear, axillary, rectal, or forehead site] in the ED or via parent report observed in the last 24h); AND
  3. Tachypnea (defined as respiratory rate (RR) above age-specific reference value) during the assessment in ED (triage or clinical examination).
* Written screening consent for participation in screening phase signed by parents/legal guardians and the patient if ≥14 years of age.

Additional inclusion criteria for intervention phase:

* Positive Mp screening test result with the Mp IgM lateral flow assay (LFA) (grade 2 or 3).
* Written informed consent for participation in intervention phase signed by parents or legal guardians and the patient if ≥14 years of age.

Exclusion criteria:

Exclusion criteria for screening phase:

• None.

Exclusion criteria for intervention phase:

* Contraindication to azithromycin: Documented allergy to azithromycin; cardiovascular disease, including bradycardia, arrhythmias, and/or QT-interval prolongation*; myasthenia gravis.

  *Co-medication with arrhythmogenic or QT-interval-prolonging drug (www.qtdrugs.org) is no exclusion criteria but will be discussed with the local investigators and/or trial management team (TMT).
* Underlying comorbidities: Cystic fibrosis or other chronic lung disorders (excluding asthma), primary or secondary immunodeficiency, sickle-cell anemia, or severe cerebral palsy.
* History of recurrent pneumonia (two or more episodes) or severe pneumonia (ICU admission or complications of CAP such as lung abscess, effusion, and empyema) in lifetime.
* Antibiotic treatment against Mp within the previous 7 days, including macrolides, tetracyclines, or fluoroquinolones.
* Referral to ICU directly from the ED.
* Inability to take oral medication.
* Parents are unlikely to reliably complete follow up (FUP) visits and questionnaires (e.g., due to language barriers or living far from the study site).

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 376 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Co-primary outcome: days to normalization of all vital signs | From enrollment until normalization of all vital signs for at least 24h assessed up to 28 days.
  Time (days) to normalization of all vital signs for at least 24h (efficacy), defined as temperature <38.0°C, respiratory rate and heart rate within age-specific reference ranges, and peripheral oxygen saturation (SpO2) on room air ≥93% assessed up to 28 days.
Co-primary outcome: community-acquired pneumonia(CAP)-related change in patient care status | From enrollment assessed up to 28 days.
  CAP-related change in patient care status within 28 days (safety), such as (re-)admission or ICU transfer assessed up to 28 days.

SECONDARY OUTCOMES:
Overall clinical outcome | From enrollment until end of treatment at 5 days.
  Overall clinical outcome based on benefits and harms (DOOR/RADAR approach) according to documentation of clinical response (normalization of all VS) and solicited adverse events (AEs) 1x/24h at the end of treatment (day 5) and each FUP visit.
Time (days) to normalization of CAP-related symptoms | From enrollment until normalization of CAP-related symptoms assessed up to 28 days.
  Time (days) to normalization of CAP-related symptoms assessed up to 28 days.
Quality of Life (QoL) Assessment assessing impact of the child's pneumonia on the family's social and health-related well-being | From enrollment assessed up to 28 days.
  QoL assessment of the patient's family with the pediatric quality of life inventory TM (PedsQLTM) family impact module and generic core scales questionnaire until day 28.
Time (days) to return to daily routine | From enrollment assessed up to 28 days.
  Time (days) to return to daily routine, defined as return to childcare/school/work of patients and their families.
Incidence of Mp-associated extrapulmonary manifestations development in patients assessed by clinical examination and/or parent report | From enrollment assessed up to 28 days.
  Development of Mp-associated extrapulmonary manifestations within 28 days after randomization based on clinical examination and/or parent report.

OTHER OUTCOMES:
Length of hospital stay (LOS) | From enrollment assessed up to 28 days.
  LOS (days) in hospitalized patients after index hospitalization.
Number of unscheduled medical visits | From enrollment assessed up to 28 days.
  Number of unscheduled medical visits (apart from the study) until day 28.
Proportion of patients (re-)treated with antibiotics for any reason | From enrollment assessed up to 28 days.
  Proportion of patients (re-)treated with antibiotics for any reason until 28 days and total antibiotic exposure in days up to 28 days.
Side effects/AEs/serious AE (SAE)s of investigational medicinal product (IMP) | From enrollment until end of treatment at 5 days.
  Side effects/AEs/SAEs of IMP.
Microbiological indicators | From enrollment assessed up to 28 days.
  Microbiological indicators (proportion of patients who cleared Mp in the upper respiratory tract (URT) within 28 days, proportion of patients in which Mp became resistant to macrolides within 28 days, proportion of patients with change in co-detecting pathogens in the URT at day 3 and 28) and inflammatory indicators (biomarker and cytokine profiling at day 3 and 28).
Other additional outcome independent of study intervention: Degree of usefulness of informational video about the study | From enrollment assessed up to 28 days.
  Degree of usefulness of informational video about the study on a five-point Likert scale. Low scores indicate a low degree of usefulness and high scores indicate a high degree of usefulness.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Berger, Prof. Dr. med., Study Chair — University Children's Hospital, Zurich
Locations (13):
- Switzerland (13):
  - Children's Hospital Aarau, Switzerland, Aarau, Canton of Aargau
  - University of Basel Children's Hospital, Switzerland, Basel, Canton of Basel-City
  - University Children's Hospital Bern, Switzerland, Bern, Canton of Bern
  - Department of Pediatrics, Fribourg Hospital, Switzerland, Fribourg, Canton of Fribourg
  - Children's Hospital of Geneva, University Hospitals of Geneva, Switzerland, Geneva, Canton of Geneva
  - Children's Hospital of Central Switzerland, Switzerland, Lucerne, Canton of Lucerne
  - Children's Hospital of Eastern Switzerland St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Department of Pediatrics, Department Mother-Woman-Child, Lausanne University Hospital, Switzerland, Lausanne, Canton of Vaud
  - Department of Pediatrics, Cantonal Hospital Winterthur, Switzerland, Winterthur, Canton of Zurich
  - University Children's Hospital Zurich, Switzerland, Zurich, Canton of Zurich
  - Department of Pediatrics, Triemli Hospital Zurich, Switzerland, Zurich, Canton of Zurich
  - Institute of Pediatrics of Southern Switzerland, EOC, Bellinzona, Switzerland, Bellinzona, Canton Ticino
  - Department of Pediatrics, Cantonal Hospital Graubuenden, Switzerland, Chur, Kanton Graubünden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meyer Sauteur PM, Krautter S, Ambroggio L, Seiler M, Paioni P, Relly C, Capaul R, Kellenberger C, Haas T, Gysin C, Bachmann LM, van Rossum AMC, Berger C. Improved Diagnostics Help to Identify Clinical Features and Biomarkers That Predict Mycoplasma pneumoniae Community-acquired Pneumonia in Children. Clin Infect Dis. 2020 Oct 23;71(7):1645-1654. doi: 10.1093/cid/ciz1059. PMID 31665253
- [Background] Meyer Sauteur PM, Truck J, van Rossum AMC, Berger C. Circulating Antibody-Secreting Cell Response During Mycoplasma pneumoniae Childhood Pneumonia. J Infect Dis. 2020 Jun 16;222(1):136-147. doi: 10.1093/infdis/jiaa062. PMID 32034406
- [Background] Meyer Sauteur PM, Seiler M, Truck J, Unger WWJ, Paioni P, Relly C, Staubli G, Haas T, Gysin C, M Bachmann L, van Rossum AMC, Berger C. Diagnosis of Mycoplasma pneumoniae Pneumonia with Measurement of Specific Antibody-Secreting Cells. Am J Respir Crit Care Med. 2019 Oct 15;200(8):1066-1069. doi: 10.1164/rccm.201904-0860LE. No abstract available. PMID 31251669
- [Background] Meyer Sauteur PM, Beeton ML; European Society of Clinical Microbiology and Infectious Diseases (ESCMID) Study Group for Mycoplasma and Chlamydia Infections (ESGMAC), and the ESGMAC Mycoplasma pneumoniae Surveillance (MAPS) study group. Mycoplasma pneumoniae: delayed re-emergence after COVID-19 pandemic restrictions. Lancet Microbe. 2024 Feb;5(2):e100-e101. doi: 10.1016/S2666-5247(23)00344-0. Epub 2023 Nov 23. No abstract available. PMID 38008103
- [Background] Kutty PK, Jain S, Taylor TH, Bramley AM, Diaz MH, Ampofo K, Arnold SR, Williams DJ, Edwards KM, McCullers JA, Pavia AT, Winchell JM, Schrag SJ, Hicks LA. Mycoplasma pneumoniae Among Children Hospitalized With Community-acquired Pneumonia. Clin Infect Dis. 2019 Jan 1;68(1):5-12. doi: 10.1093/cid/ciy419. PMID 29788037
- [Background] Williams DJ, Edwards KM, Self WH, Zhu Y, Arnold SR, McCullers JA, Ampofo K, Pavia AT, Anderson EJ, Hicks LA, Bramley AM, Jain S, Grijalva CG. Effectiveness of beta-Lactam Monotherapy vs Macrolide Combination Therapy for Children Hospitalized With Pneumonia. JAMA Pediatr. 2017 Dec 1;171(12):1184-1191. doi: 10.1001/jamapediatrics.2017.3225. PMID 29084336
- [Background] Biondi E, McCulloh R, Alverson B, Klein A, Dixon A, Ralston S. Treatment of mycoplasma pneumonia: a systematic review. Pediatrics. 2014 Jun;133(6):1081-90. doi: 10.1542/peds.2013-3729. PMID 24864174
- [Background] Gardiner SJ, Gavranich JB, Chang AB. Antibiotics for community-acquired lower respiratory tract infections secondary to Mycoplasma pneumoniae in children. Cochrane Database Syst Rev. 2015 Jan 8;1(1):CD004875. doi: 10.1002/14651858.CD004875.pub5. PMID 25566754
- [Derived] Meyer Sauteur PM, Seiler M, Tilen R, Osuna E, von Wantoch M, Sidorov S, Aebi C, Agyeman P, Barbey F, Bielicki JA, Coulon L, Deubzer B, Donas A, Heininger U, Keitel K, Kohler H, Kottanattu L, Lauener R, Niederer-Loher A, Posfay-Barbe KM, Tomaske M, Wagner N, Zimmermann P, Zucol F, von Felten S, Berger C. A randomized controlled non-inferiority trial of placebo versus macrolide antibiotics for Mycoplasma pneumoniae infection in children with community-acquired pneumonia: trial protocol for the MYTHIC Study. Trials. 2024 Oct 3;25(1):655. doi: 10.1186/s13063-024-08438-6. PMID 39363201